CLINICAL TRIAL: NCT03593018
Title: Randomized Phase 3 Study Evaluating the Efficacy and the Safety of Oral Azacitidine (CC-486) Compared to Investigator's Choice Therapy in Patient with Relapsed or Refractory Angioimmunoblastic T Cell Lymphoma
Brief Title: Efficacy and Safety of Oral Azacitidine Compared to Investigator's Choice Therapy in Patients with Relapsed or Refractory AITL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORACLE
Record Dates: First submitted 2018-07-06; First posted 2018-07-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Relapsed Angioimmunoblastic T-Cell Lymphoma; Refractory Angioimmunoblastic T-cell Lymphoma
Keywords: oral azacitidine
MeSH Terms: conditions — Immunoblastic Lymphadenopathy | interventions — Azacitidine; cc-486; romidepsin; Bendamustine Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Azacitidine (Experimental): Oral azacitidine 300mg during 14 first days of 28-days cycle for European (EU) patients, Oral azacitidine 200mg during 14 first days of 28-days cycle for Asian patients (Treatment until progression, patient decision or toxicity)
  Interventions: Drug: Oral azacitidine
- Investigator's choice therapy (Active Comparator): Romidepsin 14mg/m² on days 1, 8 and 15 of a 28-days cycle (Treatment until progression, patient decision or toxicity) or Bendamustine 120mg/m² on days 1 and 2 of a 21-days cycle (during 6 cycles) or Gemcitabine 1200mg/m² on days 1, 8 and 15 of a 28-days cycle (during 6 cycles)
  Interventions: Drug: Romidepsin; Drug: Bendamustine; Drug: Gemcitabine

INTERVENTIONS:
Drug: Oral azacitidine — Azacitidine tablets
  Other Names: CC-486
  Arms: Oral Azacitidine
Drug: Romidepsin — Romidepsin injection
  Other Names: Istodax
  Arms: Investigator's choice therapy
Drug: Bendamustine — Bendamustine injection
  Other Names: Levact
  Arms: Investigator's choice therapy
Drug: Gemcitabine — Gemcitabine injection
  Other Names: Gemzar
  Arms: Investigator's choice therapy

SUMMARY:
This study evaluates the efficacy of Oral azacitidine versus single-agent Investigator's Choice Therapy in patients with Relapsed or Refractory Angioimmunoblastic T-cell Lymphoma.

DETAILED DESCRIPTION:
Compared to B-cell Non-Hodgin Lymphoma (NHL), Angioimmunoblastic T-cell Lymphoma (AITL) is more resistant to conventional chemotherapy and is generally associated with an inferior outcome. In case of relapsed of refractory disease, survival durations are in the range of only a few months.

Several agents have been evaluated in this setting in recent years: romidepsin, bendamustine or belinostat. The response rate with these agents rarely exceeds 30% and responses are usually of limited duration.

Azacitidine is a nucleoside metabolic inhibitor indicated for the treatment of patients with various myelodysplastic syndrome (MDS) subtypes. In this case, azacitidine significantly increase the survival time compared to standard of care option. This response to azacitidine could be correlated to the existence of recurrent mutations and those mutations have also been described in AITL.

The present protocol will use Azacitidine according to the same schedule than in MDS that is continuous treatment until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all following criteria to be enrolled in the study::

1. Patient is ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Patient must understand and voluntarily sign an ICF prior to any study-specific assessments/procedures being conducted.
3. Patient is willing and able to adhere to the study visit schedule and other protocol requirements
4. Patient had local diagnosed peripheral T cell lymphoma (PTCL) with T-follicular helper (TFH) phenotype according to the criteria of the latest World Health Organization (WHO) classification based on a surgical lymph node biopsy including any one of

   * Angioimmunoblastic T cell lymphoma (AITL)
   * Follicular T cell lymphoma
   * Nodal peripheral T-cell lymphoma with TFH phenotype There should be a documented expression of minimum two TFH markers among this panel of markers : CD10, CXCL13, PD1, ICOS and BCL6 by the tumoral cells by immunohistochemistry. Biopsy at relapse or progression is not mandatory, but highly encouraged on a surgical or needle core biopsy, and diagnostic tissue should be available for central pathology review and for ancillary molecular studies.

   Local pathology report should be reviewed by the sponsor's medical monitor prior to enrollment.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3
6. Relapsed (after partial or complete response) or refractory AITL after at least one line of systemic therapy (there is no mandatory resting period after the previous treatment as long as the biochemistry and hematology labs meet the inclusion criteria as below.)
7. Meet the following lab criteria:

   * Absolute Neutrophil Count (ANC) ≥ 1,5 x 109/L (≥ 1 x 109/L if bone marrow (BM) involvement by lymphoma)
   * Platelet ≥ 75 x 109/L (≥ 50 x 109/L if BM involvement by lymphoma)
   * Hemoglobin ≥ 8 g/dL.
8. Anticipated life expectancy at least 3 months
9. At least one measurable lesion on CT that is greater than 1.5 cm in the longest diameter for nodal lesions and greater than 1.0 cm in the longest diameter for extranodal lesions. The lesion must be measurable in two perpendicular dimensions. Patients with only cutaneous disease will be excluded.
10. Female patient of childbearing potential (FCBP) may participate, providing she meets the following conditions:

    Have two negative pregnancy tests as verified by the investigator prior to starting study treatment: serum pregnancy test at Screening and negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting treatment with study treatment (Cycle 1 Day 1). She must agree to ongoing pregnancy testing during the study (before beginning each subsequent cycle of treatment), and 28 days after the last study drug administration. This applies even if the patient practices complete abstinence from heterosexual contact.

    Agrees to practice true abstinence (which must be reviewed monthly and source documented) or agrees to the use of highly effective methods of contraception from 28 days prior to starting study treatment, and must agree to continue using such precautions during study treatment (including dose interruptions) and for up to 90 days after the last study drug administration. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptom-thermal, post ovulation methods) and withdrawal are not acceptable methods of contraception. Cessation of contraception after this point should be discussed with a responsible physician.

    Agrees to abstain from breastfeeding during study participation and for at least 90 days after the last study drug administration.

    A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months).
11. Male patient must either practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agrees to avoid fathering a child, to use highly effective methods of contraception, male condom plus spermicide during sexual contact with a pregnant female or a female of childbearing potential (even if he has undergone a successful vasectomy), from starting dose of drug (cycle 1 Day 1), including dose interruptions through 90 days after receipt of the last study drug administration. Furthermore, male patient must agree to not give semen or sperm during study drug therapy and for a period of 1 year after end of study drug therapy.
12. For EU countries, patient covered by a social security system

Exclusion Criteria:

Presence of any of the following will exclude a patient from enrollment:

1. Clinical evidence of central nervous system involvement by lymphoma. Patients with suspicion of central nervous system (CNS) involvement must undergo neurologic evaluation and CT/MRI of head and lumbar puncture to exclude CNS disease.
2. Any significant medical conditions, laboratory abnormality or psychiatric illness likely to interfere with participation in this clinical study (according to the investigator's decision)
3. Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
4. Known Human Immunodeficiency Virus (HIV) or Hepatitis C Virus (HCV) infection, or evidence of positive HTLV1 serology or of active Hepatitis B (HB) Virus (HBV) infection defined as:

   * HB s Ag positive
   * HB s Ag negative, anti-HB s antibody positive and/or anti-HB c antibody positive with detectable viral DNA
5. Impaired renal function (MDRD formula or Cockcroft-Gault Creatinine Clearance < 30 ml/min) or impaired liver function tests (Serum total bilirubin level > 2.0 mg/dl [34 µmol/L] (except in case of Gilbert's Syndrome, or documented liver or pancreatic involvement by lymphoma), Serum transaminases (AST or ALT) > 3 upper normal limits) unless they are related to the lymphoma.
6. Active malignancy other than the one treated in this research. Prior history of malignancies, other than low risk MDS or chronic myelomonocytic leukemia (CMML) (with less than 5% blasts in bone marrow), unless the patient has been free of the disease for ≥ 3 years. However, patients with the following history/concurrent conditions are allowed:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histologic finding of prostate cancer (T1a or T1b) using the tumor-nodes-metastasis (TNM)] clinical staging system
   5. Early-stage gastric cancer suitable for endoscopic mucosal resection or endoscopic submucosal dissection
7. Treatment with any investigational drug within 5 half-lives before planned first cycle of study treatment and during the study. Ongoing medically significant adverse events from previous treatment, regardless of the time period.
8. Prior exposure to azacitidine and/ or any other demethylating agent (eg, decitabine)
9. Prior exposure to planned study treatment investigator's choice therapy (eg, prior exposure to gemcitabine is an exclusion if gemcitabine is the investigator's choice therapy prior to randomization)
10. Concurrent use of corticosteroids unless the patient is on a stable or decreasing dose for ≥ 1 week prior to informed consent form signature
11. Knowing or suspected hypersensitivity to active substance or to any of the excipients.
12. Pregnant, planning to become pregnant, or lactating woman
13. Candidate for hematopoietic stem cell transplantation
14. History of active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), celiac disease (ie, sprue), prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the oral azacitidine and/or predispose the patient to an increased risk of gastrointestinal toxicity per investigator's decision. Any condition causing inability to swallow tablets.
15. Significant active cardiac disease within the previous 6 months, including:

    * New York Heart Association (NYHA) class IV congestive heart failure
    * Unstable angina or angina requiring surgical or medical intervention; and/or
    * Myocardial infarction
16. Person deprived of his/her liberty by a judicial or administrative decision
17. Adult person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 18 months after first randomisation (when 18 events will occur)
  PFS using local assessment of progressive disease according to Lugano Response Criteria (2014)
Progression Free Survival (PFS) | 35 months after first randomisation (when 61 events will occur)
  PFS using local assessment of progressive disease according to Lugano Response Criteria (2014)

SECONDARY OUTCOMES:
Overall survival (OS) | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  Overall survival
PFS by the Independent Review Committee (IRC) | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  PFS by the Independent Review Committee
Overall response rate | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  Percentage of Complete Response (CR)+ Partial Response (PR) among all patients
Complete response rate (CRR) | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  Percentage of CR among all patients
Duration of response (DoR) | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  Duration of response
Time to response (TtR) | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  Time to response
PFS 2 using local assessment of progressive disease | 40 months after first randomisation (when 57 deaths will occur) or 2 years after last randomisation
  PFS 2 using local assessment of progressive disease
Quality of Life Questionnaire (QLQ-C30) | 2 years after last randomisation
  questionnaire at baseline and at least one follow-up
Number of Serious Adverse Events (SAE) | 2 years after last randomisation
  Treatment discontinuation, adverse events, deaths

CONTACTS AND LOCATIONS:
Overall Officials: Jehan DUPUIS, MD, Study Chair — Henri Mondor University Hospital; François LEMONNIER, MD, Study Chair — Henri Mondor University Hospital; Kunihiro TSUKASAKI, MD, Study Chair — Saitama Medical University International Medical Center
Locations (27):
- Austria (2):
  - University Hospital for Internal Medicine - University Hospital Graz, Graz
  - Medical University of Vienna, Vienna
- Belgium (3):
  - A. Z. Sint-Jan Brugge-Oostende AV, Bruges
  - Cliniques Universitaires de Bruxelles - Hôpital Erasme, Brussels
  - CHU UCL Namur - Site Godinne, Yvoir
- Aarhus University Hospital, Aarhus, Denmark
- France (17):
  - Institut d'Hématologie de Basse Normandie, Caen
  - CHU de Clermont-Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital Necker, Paris
  - Hôpital Saint-Louis, Paris
  - CHU Haut-Lévèque - Centre François Magendie, Pessac
  - CHU Lyon-Sud, Pierre-Bénite
  - CH Annecy Genevois, Pringy
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - IUCT - Oncopole, Toulouse
  - CHRU de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
- United Kingdom (4):
  - University College London Hospital, London
  - The Christie, Manchester
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupuis J, Bachy E, Morschhauser F, Cartron G, Fukuhara N, Daguindau N, Casasnovas RO, Snauwaert S, Gressin R, Fox CP, d'Amore FA, Staber PB, Tournilhac O, Bouabdallah K, Thieblemont C, Andre M, Rai S, Ennishi D, Gkasiamis A, Nishio M, Fornecker LM, Delfau-Larue MH, Sako N, Mule S, de Leval L, Gaulard P, Tsukasaki K, Lemonnier F. Oral azacitidine compared with standard therapy in patients with relapsed or refractory follicular helper T-cell lymphoma (ORACLE): an open-label randomised, phase 3 study. Lancet Haematol. 2024 Jun;11(6):e406-e414. doi: 10.1016/S2352-3026(24)00102-9. PMID 38796193
- See also: Website of The Lymphoma Study Research Organisation (LYSARC) — https://www.lysarc.org/